CLINICAL TRIAL: NCT07216196
Title: The Effect of Dyadic Metacognitive Strategy Training in Autistic Youth or Young Adults and a Primary Caregiver
Brief Title: The Feasibility of a Remote Problem-Solving Intervention for Autistic Adolescents or Young Adults and a Caregiver
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Missouri-Columbia (Other)
Responsible Party: Principal Investigator, Melanie Tkach, Assistant Professor, University of Missouri-Columbia
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Treatment
Other Study IDs: 2126948
Record Dates: First submitted 2025-10-09; First posted 2025-10-14 (Actual); Last update posted 2026-01-30 (Actual); Status verified 2026-01

CONDITIONS: Autism
Keywords: Occupational Therapy; Autism; Transition to Adulthood; Waitlist Crossover
MeSH Terms: conditions — Autistic Disorder | interventions — Health Resources

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Remote Metacognitive Strategy Training (Experimental): The intervention group will complete the remote metacognitive strategy training intervention immediately.
  Interventions: Behavioral: Pathways and Resources for Engagement and Participation (PREP)
- Waitlist Control (No Intervention): The waitlist control group will wait 12 weeks without intervention. Then, they will crossover into the intervention arm and receive the remote metacognitive strategy training intervention.

INTERVENTIONS:
Behavioral: Pathways and Resources for Engagement and Participation (PREP) — Pathways and Resources for Engagement and Participation (PREP) is a collaborative problem-solving intervention that targets environmental barriers-physical, social, attitudinal, familial, and institutional-while leveraging adolescent and family strengths. Caregivers are integrated as key supports. The five-step process includes: (1) make goals, (2) map out a plan, (3) make it happen, (4) measure outcomes, and (5) move forward. We will set four activity-based transition goals using the Transition Planning Inventory-2nd Edition and Goal Attainment Scaling. Providers will use guided discovery to help adolescents and caregivers identify strategies that modify activities or environments to support participation in transition activities. Adolescents and caregivers will implement strategies between sessions and revise strategies with the provider in future sessions if unsuccessful. Participants will complete 12 weekly 60-min remote PREP sessions over 12-16 weeks.
  Arms: Remote Metacognitive Strategy Training

SUMMARY:
This project seeks to evaluate the feasibility and acceptability of a remote metacognitive strategy training intervention in transition-age autistic adolescents and young adults and a primary caregiver. We will also conduct limited efficacy testing.

DETAILED DESCRIPTION:
The U.S. healthcare and educations systems are failing autistic adolescents and young adults (AYAs) through inadequate or inaccessible services that hinder the development of independent living skills for long-term participation, health, and the transition to adulthood. In fact, only 19% of autistic AYAs who received special education services live independently and just over half were employed by their early 20s. These trends negatively impact autistic people's health and well-being and result in substantial familial and societal costs ranging from $1.4 to $2.4 million per person. Existing rehabilitation interventions for autistic AYAs primarily target isolated skills and overlook caregiver influences on AYA outcomes, so intervention gains do not translate to improvements in long-term participation or transition outcomes.

Pathways and Resources for Engagement and Participation (PREP), an MCST intervention for AYAs with physical disabilities and their families, may improve participation, health, and transition outcomes in autistic youths. PREP is a problem-solving approach to family-chosen goals that focuses on activity or environmental modifications over skill development. PREP improves activity performance and participation in AYAs with physical disabilities and autistic children ages 6-12. However, PREP has not been rigorously tested with autistic AYAs and caregivers. The critical next step is to test whether PREP improves participation, health and well-being, and transition outcomes in autistic AYAs. The overall study hypothesis is that PREP will be feasible for autistic AYAs and caregivers.

We will conduct a randomized controlled trial with waitlist crossover in autistic AYAs and their caregivers (e.g., youth-caregiver dyads). Youth-caregiver dyads will include one autistic AYA and one primary caregiver that meet other study inclusion criteria and provide electronic informed consent and assent. AYA-caregiver dyads will complete a baseline assessment (T1) of AYA activity performance, participation, and mental health. Then, they will be randomly assigned to intervention or waitlist control groups. The intervention group will complete remote PREP immediately (one hour/week x 12 weeks), and the waitlist control group will wait 12 weeks without intervention and then complete remote PREP (one hour/week x 12 weeks). The intervention group will complete post-intervention (T2) and follow-up (T3) assessments. The waitlist control group will complete second baseline (T2) and post-intervention (T3) assessments. AYA-caregiver dyads will complete one in-depth, semi-structured interview post-intervention to determine intervention acceptability.

We aim to test the feasibility of remote PREP for autistic AYAs and their caregivers. We hypothesize that feasibility data (e.g., recruitment, retention, and intervention adherence) will indicate that the study protocol and intervention can be implemented with autistic AYAs and a primary caregiver. We also hypothesize that acceptability data will indicate adequate intervention acceptability and inform optimization for future trials. Our second aim is to conduct limited efficacy testing to identify the preliminary effect of remote PREP on AYA outcomes. We hypothesize that effect size estimations will indicate the remote PREP has a greater positive effect, compared to waitlist control, on AYA activity performance, participation, health, and transition outcomes.

ELIGIBILITY:
Inclusion Criteria:

* Autistic adolescents aged 13-21 AND one primary parent, guardian, or caregiver aged 18 or older
* At least one year remaining in high school
* Ability to engage in reciprocal conversation
* Ability to provide informed consent/assent as part of an adapted procedure designed to prevent coercion and protect the rights of autistic adolescents with or without intellectual disability

Exclusion Criteria:

* Severe or profound intellectual disability (IQ<35)
* Severe mental health conditions that interfere with ability to participate in the intervention
* Currently enrolled in community-based transition services redundant with remote PREP

Ages: 13 Years to 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 24 (Estimated)
Dates: Start 2026-02-01 (Estimated); Primary Completion 2026-11-03 (Estimated); Study Completion 2027-05-03 (Estimated)

PRIMARY OUTCOMES:
Acceptability of Intervention Measure (AIM) | Intervention - week 13; Waitlist control - week 25
  Measure of intervention acceptability. Self-report Likert scale from 1 -completely disagree to 5 - completely agree
Semi-Structured Interview | Intervention - week 13; Waitlist control - week 25
  A brief interview to gather participant perceptions of the intervention, including their perceived benefit and practicality of the intervention and suggestions for improvement for the intervention. Data will be qualitative interview transcripts.

SECONDARY OUTCOMES:
Participation and Environment Measure - Child and Youth | Intervention - Baseline (week 0), post-intervention (week 13), follow-up (week 25); Waitlist control- Baseline (week 0), second baseline (week 13), post-intervention (week 25)
  Caregiver proxy report measure of adolescent activity participation at home, school, and in the community. Caregivers rate adolescents' participation frequency (0 - never to 7 - daily) and involvement (1 - minimally involved to 5 - very involved). Higher scores represent better adolescent participation.
Youth, Young Adult Participation and Environment Measure | Intervention - Baseline (week 0), post-intervention (week 13), follow-up (week 25); Waitlist Control - Baseline (week 0), second baseline (week 13), post-intervention (week 25)
  Self-report measure of adolescent and young adult activity participation at home, school, and in the community. Adolescents and young adults rate their participation frequency (0 - never to 7 - daily) and involvement (1 - minimally involved to 5 - very involved). Higher scores represent better adolescent participation.
Patient-Reported Outcomes Measurement Information System Pediatric Global Health Measure 7+2 | Baseline (week 0), post-intervention (week 13), follow-up (week 25); Baseline (week 0), second baseline (week 13), post-intervention (week 25)
  Informant and self-report questionnaire of adolescent and young adult physical and mental health. Item responses range from 1 - poor to 5 - excellent. Higher scores represent better health.
Transition Readiness Scale | Intervention - Baseline (week 0), post-intervention (week 13), follow-up (week 25); Waitlist Control - Baseline (week 0), second baseline (week 13), post-intervention (week 25)
  Informant and self-report measure of adolescent transition readiness (education, work, independent living). Self-report scale that ranges from 1 - not true for me/my child to 4 - true for me/my child. Higher scores represent better transition readiness.
Canadian Occupational Performance Measure (COPM) | Intervention - Baseline (week 0), post-intervention (week 13), follow-up (week 25); Waitlist control- Baseline (week 0), second baseline (week 13), post-intervention (week 25)
  Self-report measure of activity performance. Minimum = 1, Maximum = 10. Higher scores mean better performance.

OTHER OUTCOMES:
Transition Planning Inventory - 3rd Edition | Baseline (Week 0)
  A four-section survey about student preferences and interests for post-secondary outcomes. Respondents identify a goal for work, school, or independent living and answer five open-ended questions related to their goal. Qualitative responses will be used to co-create goals for intervention sessions.

CONTACTS AND LOCATIONS:
Overall Officials: Melanie M. Tkach, PhD, Principal Investigator — University of Missouri-Columbia
Locations (1):
- University of Missouri - Columbia, Columbia, Missouri, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Anderson KA, Sosnowy C, Kuo AA, Shattuck PT. Transition of Individuals With Autism to Adulthood: A Review of Qualitative Studies. Pediatrics. 2018 Apr;141(Suppl 4):S318-S327. doi: 10.1542/peds.2016-4300I. PMID 29610413
- [Background] Fujiwara T, Takanashi Y, Nakae S, Tsutsui T, Fukuchi S, Ogoshi T, Endo M, Hashimoto A, Hayashi H, Koyanagi H. [Clinical results of the intra-aortic balloon pumping after cardiac surgery (author's transl)]. Kyobu Geka. 1981 Jul;34(7):497-503. No abstract available. Japanese. PMID 7311242
- [Background] Kang LJ, Huang HH, Wu YT, Chen CL. Initial evaluation of an environment-based intervention for participation of autistic children: a randomized controlled trial. Disabil Rehabil. 2024 May;46(9):1851-1861. doi: 10.1080/09638288.2023.2209743. Epub 2023 May 15. PMID 37183406
- [Background] Hsieh YH, Ryan M, Anaby D. Towards multi-faceted outcomes of participation-based interventions: mapping the PREP's effects for children and youth with disabilities. Disabil Rehabil. 2024 Oct;46(20):4825-4834. doi: 10.1080/09638288.2023.2280084. Epub 2023 Nov 21. PMID 39319861
- [Background] Little LM, Cohen SR, Tomchek SD, Baker A, Wallisch A, Dean E. Interventions to Support Social Participation for Autistic Children and Adolescents in Homes and Communities (2013-2021). Am J Occup Ther. 2023 Mar 1;77(Suppl 1):7710393200. doi: 10.5014/ajot.2023.77S10020. PMID 37611261
- [Background] Baker A, Tomchek SD, Little LM, Wallisch A, Dean E. Interventions to Support Participation in Basic and Instrumental Activities of Daily Living for Autistic Children and Adolescents (2013-2021). Am J Occup Ther. 2023 Mar 1;77(Suppl 1):7710393140. doi: 10.5014/ajot.2023.77S10014. PMID 37562056
- [Background] Egilson ST, Jakobsdottir G, Olafsson K, Leosdottir T. Community participation and environment of children with and without autism spectrum disorder: parent perspectives. Scand J Occup Ther. 2017 May;24(3):187-196. doi: 10.1080/11038128.2016.1198419. Epub 2016 Jun 22. PMID 27329683
- See also: PREP Intervention Protocol — https://canchild.ca/shop/25-prep-intervention-protocol/